CLINICAL TRIAL: NCT00551590
Title: A Randomized, Placebo-Controlled, 4-period, Crossover Study to Assess the Impact of MK-0431 (Sitagliptin) on Incretin Effect and the Role of Specific Incretin Hormones in Patients With Type 2 Diabetes Mellitus
Brief Title: Effect of Sitagliptin on Incretin Effect in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Joerg Schirra, Prof. Dr. med., Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: SITEX-02; EudraCT 2007-001050-83
Record Dates: First submitted 2007-10-30; First posted 2007-10-31 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes mellitus; DPP-4 inhibitor; sitagliptin; exendin(9-39); GLP-1
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Sitagliptin Phosphate; exendin (9-39)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Placebo Comparator): placebo PO (placebo control for sitagliptin) for three days. Saline IV (placebo control for exendin(9-39) on two consecutive study days.
  Interventions: Drug: Placebo tablet; Drug: Saline infusion
- 2 (Experimental): Sitagliptin 100 mg PO for three days. Saline IV (placebo control for exendin(9-39)) on two consecutive study days
  Interventions: Drug: Sitagliptin tablet; Drug: Saline infusion
- 3 (Experimental): Sitagliptin 100 mg PO for three days. Exendin(9-39) IV on two consecutive study days.
  Interventions: Drug: Sitagliptin tablet; Drug: Exendin(9-39) infusion
- 4 (Placebo Comparator): placebo PO (placebo control for sitagliptin) for three days. Exendin(9-39)IV on two consecutive study days.
  Interventions: Drug: Placebo tablet; Drug: Exendin(9-39) infusion

INTERVENTIONS:
Drug: Placebo tablet — placebo PO (placebo control for sitagliptin) for three days
  Arms: 1; 4
Drug: Sitagliptin tablet — Sitagliptin 100 mg PO for three days.
  Arms: 2; 3
Drug: Saline infusion — Saline IV (placebo control for exendin(9-39)) on two consecutive study days
  Arms: 1; 2
Drug: Exendin(9-39) infusion — Exendin(9-39) IV on two consecutive study days.
  Arms: 3; 4

SUMMARY:
The purpose of this study is to assess the effect of the DPP-4 inhibitor sitagliptin on the incretin effect in patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Following a meal, gut-produced incretin hormones such as glucagon-like peptide-1 (GLP-1) and glucose-dependent insulinotropic polypeptide (GIP) are released into the circulation. Because GLP-1 and GIP mediate grossly 60% of the insulin-stimulatory action, the so-called incretin effect, both are crucial components of a natural endogenous system guaranteeing glucose homeostasis. In addition, GLP-1 lowers glucagon secretion from pancreatic alpha-cells and delays nutrient delivery from the stomach by inhibiting gastric emptying. The rise in insulin concentration enhances glucose clearance in peripheral tissues such as muscle, and the lower glucagon concentration combined with the rise in insulin reduces hepatic glucose production. By enhancing glucose clearance and lowering hepatic glucose production, the post-meal glucose excursion is reduced.

Both GLP-1 and GIP are degraded by the enzyme dipeptidylpeptidase-4 (DPP-4). Inhibition of DPP-4 by the specific DPP-4 inhibitor Sitagliptin increases plasma levels of both GLP-1 and GIP, and reduces postprandial glycemia.

Although important in healthy subjects, the role of the incretin hormones in patients with T2DM is unclear. In T2DM the insulinotropic efficacy of GIP is reduced and the postprandial release of GLP-1 is diminished.

Therefore, the aim of this study in T2DM is to quantify the incretin effect with and without the DPP-4 inhibitor sitagliptin. The specific GLP-1 receptor antagonist exendin(9-39) will be used to quantify the contribution of both GLP-1 and GIP to the incretin effect in patients with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Women with T2DM without childbearing potential
* Male patients with T2DM using a double-barrier method of contraception
* must be able to complete a 1 week wash-out of current anti-diabetic medications (patients on PPARγ must be off for at least 4 weeks)
* no medications which may alter gastric motility (i.e. acetaminophen, erythromycin) except for cardiac medication at a stable dose.
* Age 30-70 years
* HbA1c ≤9% at screening
* BMI<40 kg/m2
* Must have a fasting blood glucose of ≤11.1 mmol/L (200 mg/dL) at screening
* Able to provide written informed consent prior to study participation
* Able to communicate well with the investigator and comply with the requirements of the study
* Able to maintain dietetic restrictions and to perform measurements of blood glucose on a daily basis (fasting and two-hours postprandial). Patients must be informed the investigator if fasting glucose is above 200mg/dl or two hours postprandially blood glucose concentration above 240mg/dl is being measured.

Exclusion Criteria:

* T1DM, diabetes as a result of pancreatic injury, or secondary forms of diabetes (eg. Cushing, acromegaly)
* Females with childbearing potential, breastfeeding and pregnant women
* Need for insulin within the previous 3 months
* Use of Thiazolidinediones in the previous 4 weeks
* Significant concomitant disease or complications of diabetes (i.e. nephropathy, autonomic dysfunction, orthostasis).
* Fasting triglycerides >5.1 mmol/L (>450 mg/dL) within the past 4 weeks.
* Treatment with systemic steroids and thyroid hormone (unstable dosage).
* Patients with any history of gastrointestinal surgery, e.g. partial bowel resections, partial gastric resections, etc.
* Participation in any clinical investigation within 4 weeks prior to dosing or longer if required by local regulation.
* Donation or loss of 400 mL or more of blood within 8 weeks prior to dosing.
* Significant illness within the two weeks prior to dosing.
* Past medical history of clinically significant ECG abnormalities or a family history of a prolonged QT-interval syndrome.
* History of clinically significant drug allergy; history of atopic allergy (asthma, urticaria, eczematous dermatitis). A known hypersensitivity to the study drug or drugs similar to the study drug.
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs or which may jeopardize the subject in case of participation in the study. The investigator should be guided by evidence of any of the following:

  * history of inflammatory bowel syndrome, gastritis, ulcers, gastrointestinal or rectal bleeding;
  * history of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection;
  * history or clinical evidence of pancreatic injury or pancreatitis;
  * history or presence of impaired renal function as indicated by abnormal creatinine or urea val-ues or abnormal urinary constituents (e.g., albuminuria);
  * evidence of urinary obstruction or difficulty in voiding at screening;
* Polymorphonuclears <1500/µL at inclusion or platelet count < 100,000/μL at screening and base-line.
* History of immunocompromise.
* Evidence of liver disease as indicated by abnormal liver function tests such as SGOT, SGPT, GGT, alkaline phosphatase, or serum bilirubin. SGOT, SGPT, GGT and alkaline phosphatase must not exceed twice the upper limit of the normal range, and serum bilirubin should not exceed the value of 27 µmol/L (1.6 mg/dL).
* History of drug or alcohol abuse within the 12 months prior to dosing or evidence of such abuse as indicated by the laboratory assays conducted during the screening evaluations.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-12; Primary Completion 2008-12 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To asses the effect of sitagliptin compared to placebo and to coadministration of sitagliptin and the GLP-1 receptor antagonist exendin(9-39)NH2 on the incretin effect after an oral glucose challenge. | during 240 minutes after ingestion of an OGTT

SECONDARY OUTCOMES:
Plasma glucagon, plasma GIP, plasma GLP-1, Insulin, C-peptide, plasma glucose profiles. 13CO2 exhalation kinetics assessing gastric emptying | during 240 minutes after ingestion of an OGTT

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Schirra, MD, Principal Investigator — Clinical Research Unit, Dept. of Internal Medicine II, University of Munich
Locations (1):
- Clinical Research unit, Dept. of Internal Medicine II - Großhadern, University of Munich, Munich, Germany

REFERENCES:
- [Background] Schirra J, Sturm K, Leicht P, Arnold R, Goke B, Katschinski M. Exendin(9-39)amide is an antagonist of glucagon-like peptide-1(7-36)amide in humans. J Clin Invest. 1998 Apr 1;101(7):1421-30. doi: 10.1172/JCI1349. PMID 9525985
- [Background] Schirra J, Nicolaus M, Roggel R, Katschinski M, Storr M, Woerle HJ, Goke B. Endogenous glucagon-like peptide 1 controls endocrine pancreatic secretion and antro-pyloro-duodenal motility in humans. Gut. 2006 Feb;55(2):243-51. doi: 10.1136/gut.2004.059741. Epub 2005 Jun 28. PMID 15985560
- [Background] Nauck M, Stockmann F, Ebert R, Creutzfeldt W. Reduced incretin effect in type 2 (non-insulin-dependent) diabetes. Diabetologia. 1986 Jan;29(1):46-52. doi: 10.1007/BF02427280. PMID 3514343
- [Derived] Aulinger BA, Bedorf A, Kutscherauer G, de Heer J, Holst JJ, Goke B, Schirra J. Defining the role of GLP-1 in the enteroinsulinar axis in type 2 diabetes using DPP-4 inhibition and GLP-1 receptor blockade. Diabetes. 2014 Mar;63(3):1079-92. doi: 10.2337/db13-1455. Epub 2013 Dec 2. PMID 24296715